CLINICAL TRIAL: NCT03412448
Title: The Prevalence of Chronic Pain and Continued Opioid Use After Cardiac
Brief Title: The Prevalence of Chronic Pain and Continued Opioid Use After Cardiac Surgery
Acronym: Doul-Card
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-2188
Record Dates: First submitted 2018-01-19; First posted 2018-01-26 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Chronic Pain; Cardiac Surgery; Opioid Use
Keywords: chronic pain; cardiac surgery; opioids
MeSH Terms: conditions — Chronic Pain | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observation — Observation,

SUMMARY:
The authors propose to evaluate the prevalence of chronic post-operative pain (CPOP) and continued opioid use in the population that has undergone cardiac surgery at the Montreal Heart Institute. In addition, the authors wish to evaluate the presence of known risk factors for CPOP in this population.

DETAILED DESCRIPTION:
This study will use a 15-minute telephone survey to prospectively evaluate the prevalence and intensity of chronic pain 6 months and 1 year after cardiac surgery. Data on the level of post-operative pain experienced on days 1 to 4, at the time of surgery, as well as opioid consumption, adjuvant pain treatments and other variables of interest that are currently recorded prospectively at time of surgery will be culled from patient charts. Additionally, the possibility of continued opioid use by patients at 6 months post-surgery will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

All patients who have surgery at the Montreal Heart Institute between October 1 2017 and October 1 2018 will be eligible for selection.

Exclusion Criteria:

Patients who have declined to be contacted after surgery as noted on the MHI form "Consent for futur projects".

All patients who accepted to be contacted but decline to participate when contacted after their surgery.

Patients who cannot be reached by phone. Patients who cannot speak French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: population that has undergone cardiac surgery at the MHI.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-06-15 (Estimated); Study Completion 2018-08-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of CPOP | 6 (+ or - two weeks) months after surgery
  Prevalence of CPOP at 6-months post-surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
Data will not be shared

REFERENCES:
- [Background] Choiniere M, Watt-Watson J. Persistent postoperative nonanginal pain after cardiac surgery. CMAJ. 2014 Aug 5;186(11):855. doi: 10.1503/cmaj.114-0057. No abstract available. PMID 25097223
- [Background] Alam A, Gomes T, Zheng H, Mamdani MM, Juurlink DN, Bell CM. Long-term analgesic use after low-risk surgery: a retrospective cohort study. Arch Intern Med. 2012 Mar 12;172(5):425-30. doi: 10.1001/archinternmed.2011.1827. PMID 22412106
- [Background] Mazzeffi M, Khelemsky Y. Poststernotomy pain: a clinical review. J Cardiothorac Vasc Anesth. 2011 Dec;25(6):1163-78. doi: 10.1053/j.jvca.2011.08.001. Epub 2011 Sep 29. No abstract available. PMID 21955825